CLINICAL TRIAL: NCT04777942
Title: Neoadjuvant Transartery Chemoembolization Plus Artery Infusion Chemotherapy With Surgery Versus Surgery Alone for Hepatocellular Carcinoma Patients With High-risk Barcelona Clinic Liver Cancer (BCLC) A Stage: a Randomized Clinical Trial
Brief Title: Neo-TACE-HAIC for High-risk BCLC A Stage HCC (NeoconceptA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2020-322
Record Dates: First submitted 2021-02-28; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neo-TACE-HAIC with surgery (Experimental): transartery chemoembolization with lipiodol and EADM, FOLFOX (Oxa 85mg/m2 2h+CF 400mg/m2 2h+5FU 400mg/m2 10min+5FU 1200mg/m2 23h)-based artery infusion chemotherapy, followed by hepatic resection
  Interventions: Procedure: neo-TACE-HAIC+Surgery
- surgery alone (Active Comparator): hepatic resection remove the liver tumors
  Interventions: Procedure: Surgery alone

INTERVENTIONS:
Procedure: neo-TACE-HAIC+Surgery — transartery chemoembolization with lipiodol and EADM, FOLFOX (Oxa 85mg/m2 2h+CF 400mg/m2 2h +5FU 400mg/m2 10min+5FU 1200mg/m2 23h)-based artery infusion chemotherapy, followed by hepatic resection
  Arms: neo-TACE-HAIC with surgery
Procedure: Surgery alone — hepatic resection remove the liver tumors
  Arms: surgery alone

SUMMARY:
Hepatocellular carcinoma (HCC) patients is a common disease in the East Asia. Although resection was recommend for early stage (BCLC A stage) patients according to the BCLC (Barcelona clinical liver cancer) system, increasing studies suggested that preoperative transarterial therapy may decrease the recurrence risk for those with high-risk factors. However, the clinical value is still undertermined. Recently, FOLFOX (Oxaliplatin and 5-fluorouracil) based hepatic artery infusion chemotherapy (HAIC) exhibited high response rate for unresectable HCC. Pilot study showed TACE combined HAIC (TACE-HAIC) had better tumor response, with low progression disease rate. Whether TACE-HAIC would improve survival for BCLC A stage patients with high-risk factors is need to further to study. A randomized clinical trial compared neo-TACE-HAIC with surgery versus surgery alone is aimed to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years;
* BCLC A stage with high-recurrence risk factor;
* Patients with resectable primary hepatocellular carcinoma;
* Child-Pugh A or B (7 score) liver function;
* The volume of residual liver more than 30%

Exclusion Criteria:

* • With unresectable HCC

  * Pregnant woman or sucking period;
  * With other malignant cancer;
  * Received anti-HCC therapy before this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival, PFS | 36 months
  PFS was calculated from the date of starting treatment to the date of progression, of disease or death

SECONDARY OUTCOMES:
Overall survival, OS | 60 months
  OS was calculated from the date of starting treatment to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No